CLINICAL TRIAL: NCT00521274
Title: A Phase II Trial to Assess the Activity of MVA 5T4 (Trovax®) Plus Docetaxel Versus Docetaxel Alone in Patients With Progressive Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Study of Trovax® Plus Docetaxel Versus Docetaxel Alone in Patients With Progressive Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Oxford BioMedica halted TroVax injections
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#0407-0036; PCa-07-101 (Other: Principal Investigator)
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Progressive Hormone Refractory Prostate Cancer; HRPC; MVA 5T4; Trovax®; Docetaxel; M3thodist
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TroVax; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients randomized to Arm 1 will receive treatment cycles of Docetaxel and vaccine.
  PI relocated, data not available.
  Interventions: Biological: MVA 5T4
- 2 (Active Comparator): Patients randomized to Arm 2 will receive Docetaxel 75 mg/m2 on Day 1 of each cycle (1 cycle = 3 weeks). Patients who demonstrate disease progression will continue with their chemo as scheduled in Arm 2 but will also begin to receive TroVax® (cross-over).
  PI relocated, data not available.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: MVA 5T4 — Docetaxel will be administered at the completion of the first three TroVax® injections. Patients will receive Docetaxel 75 mg/m2 on Day 1 of each cycle (1 cycle = 3 weeks). Patients will receive up to 10 total Docetaxel infusions over the course of the study. Subsequent TroVax® injections will be delivered on Day 1 of each Docetaxel cycle, 2 hours prior to the chemotherapy administration.
  Other Names: TroVax
  Arms: 1
Drug: Docetaxel — Patients will receive Docetaxel 75 mg/m2 on Day 1 of each cycle (1 cycle = 3 weeks). Patients who demonstrate disease progression will continue with their chemo as scheduled in Arm 2 but will also begin to receive TroVax® (cross-over). Patients will receive up to 10 total Docetaxel infusions over the course of the study. If patients cross-over, TroVax® will be administered 2 hours prior to the chemotherapy administration.
  Other Names: Taxotere
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the role of combination therapy with Trovax plus Docetaxel or Docetaxel alone in patients with prostate cancer with a rising prostate specific antigen (PSA).

DETAILED DESCRIPTION:
Docetaxel is the most active chemotherapeutic agent in the treatment of prostate cancer.

Trovax is vaccine that targets 5T4 receptors on tumor cells. 5T4 has been detected in the majority of primary prostate cancers. Based on pre-clinical and clinical data, it may be advantageous to administer a cancer vaccine before chemotherapy to enhance immune responses, thus leading to a more therapeutic approach for patients with metastatic androgen independent prostate cancer (AIPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Progressive disease after androgen deprivation.
* ECOG Status < 2.
* No prior chemotherapy for prostate cancer therapy
* At least four weeks have lapsed since prior chemotherapy (if administered)
* Patients on stable doses of bisphosphonates that show subsequent tumor progression may continue on this medication; however, patients are not allowed to initiate bisphosphonate therapy within one month prior to starting therapy or throughout the study.
* Clinically immunocompetent.
* Free of clinically apparent/active autoimmune disease
* Absolute Lymphocyte Count ≥ 500/µl, ANC >1200/µl, Platelet count >100,000/µl, Hemoglobin > 10 mg/dl, Peripheral neuropathy <1.
* No evidence of active ischemia on ECG
* Age greater 18 years

Exclusion Criteria:

* Patients who have received prior chemotherapy.
* Patients receiving any other hormonal therapy, including any dose of megestrolacetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid must discontinue the agent for at least 4 weeks prior to enrollment. Progressive disease (as defined above) must be documented after discontinuation of the hormonal therapy.
* Patients that initiate bisphosphonate therapy within one month prior to starting therapy or throughout the study.
* No supplements or complementary medicines/botanicals are permitted during the study, except for any combination of the following: conventional multivitamin supplements, selenium, lycopene, soy supplements, Vitamin E
* Patients should review the label with their doctor prior to enrollment, and discontinue disallowed agents prior to study enrollment
* Major surgery or radiation therapy completed < 4 weeks prior to enrollment.
* Prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.
* "Currently active" second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy more than 5 years previously and have no known evidence of residual or recurrent disease
* Serious intercurrent infections or nonmalignant medical illnesses which are uncontrolled.
* Psychiatric illnesses/social situations that would limit compliance with protocol requirements.
* AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used. The bilirubin must be within normal limits.
* Renal function creatinine ≥1.5 x ULN.
* Known allergy to egg proteins.
* Known allergy to neomycin.
* History of allergic response to previous vaccinia vaccinations.
* Chronic oral corticosteroid use (especially anti-emetics) unless prescribed as replacement therapy in the case of adrenal insufficiency.
* Known to test positive for HIV or hepatitis B or C - testing prior to study not required.
* Clinical indication of reduced cardiac function or an ejection fraction of ≤ 40%.
* Requirement for radiotherapy (this is a sign of disease progression and is classed as a withdrawal criterion).
* Concurrent chemotherapy, immunotherapy and radiation therapy
* No investigational or commercial agents or therapies other than those included in protocol treatment may be administered with the intent to treat the patient's malignancy.
* Prior exposure to TroVax®.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to PSA progression Safety: To compare adverse events, laboratory measurements and vital sign measurements between the treatment groups | PSA measured every 6 weeks

SECONDARY OUTCOMES:
PSA response rate Tumor response Overall survival | PSA and tumor response measured every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No